CLINICAL TRIAL: NCT00529269
Title: Patient Reported Outcomes in Renal Transplant Patients With and Without Gastrointestinal Symptoms
Brief Title: Measurement of Patient Reported Outcomes in Korean Renal Transplant Patients With and Without Gastrointestinal (GI) Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CERL080AKR03
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Renal Transplant
Keywords: Renal Transplant Patients, GI symptom, Enteric-coated mycophenolate sodium

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
This study will evaluate the impact that GI complaints have on patient-reported outcomes and to determine if there is improvement in patient-reported outcomes when converted from mycophenolate mofetil (MMF) to Enteric-coated mycophenolate sodium (EC-MPS)

ELIGIBILITY:
Inclusion Criteria:

* Received kidney transplant at least 1 month prior to study enrollment
* Receiving immunosuppressive regimen that includes MMF for at least 2 weeks prior to study enrollment
* Eligible to convert to enteric-coated mycophenolate sodium (EC-MPS) because of GI complaints OR not currently experiencing GI complaints and stable on current immunosuppressive regimen
* At least 18 years of age
* Willing to provide written informed consent
* Able to meet all study requirements including completing electronically-administered questionnaires and completing two study visits.

Exclusion Criteria:

* GI symptoms assumed or known not to be caused by MPA (Mycophenolic acid) therapy (e.g. oral biphosphonates induced, infectious diarrhea)
* Acute rejection < 1 week prior to study enrollment
* Woman of child-bearing potential who is planning to become pregnant or is pregnant and/or lactating who is unwilling to use effective means of contraception
* Presence of psychiatric illness (i.e., schizophrenia, major depression) that, in the opinion of the site investigator, would interfere with study requirements;
* Undergoing acute medical intervention or hospitalization
* Any other medical condition that, in the opinion of the site investigator based on recall or chart review, would interfere with completing the study, including but not limited to, visual problems or cognitive impairment
* Receiving any investigational drug or have received any investigational drug within 30 days prior to study enrollment.

Other protocol-defined inclusion /exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Symptom severity is assessed by the GSRS (GI Symptom Rating Scale); Health-related Quality of Life (HRQL) is assessed by the GIQLI (GI Quality of Life) Index.

SECONDARY OUTCOMES:
Impact of immunosuppressive-induced GI symptoms on patient's perception of symptom severity and HRQL.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Chair — Novartis
Locations (2):
- South Korea (2):
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul

REFERENCES:
- [Background] Hwang HS, Hyoung BJ, Kim S, Oh HY, Kim YS, Kim JK, Kim YH, Kim YL, Kim CD, Shin GT, Yang CW. Improved gastrointestinal symptoms and quality of life after conversion from mycophenolate mofetil to enteric-coated mycophenolate sodium in renal transplant patients receiving tacrolimus. J Korean Med Sci. 2010 Dec;25(12):1759-65. doi: 10.3346/jkms.2010.25.12.1759. Epub 2010 Nov 24. PMID 21165291